CLINICAL TRIAL: NCT00733538
Title: Stage I Multiple Myeloma Treatment
Acronym: IFM-01-04
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de Nice (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Treatment
Other Study IDs: IFM-04-01
Record Dates: First submitted 2008-08-12; First posted 2008-08-13 (Estimated); Last update posted 2024-04-12 (Actual); Status verified 2009-02

CONDITIONS: Multiple Myeloma
Keywords: stage I multiple myeloma
MeSH Terms: conditions — Multiple Myeloma | interventions — Zoledronic Acid

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Active Comparator): patients receiving zometa treatment
  Interventions: Drug: zometa
- 2 (No Intervention): No treatment, just follow-up

INTERVENTIONS:
Drug: zometa — patients receiving treatment during their follow-up
  Arms: 1

SUMMARY:
* Assessment of survival without progression of stage I MM in two groups: arm A: simple survey and arm B: administration of Zoledronate.
* Describe different progression's type noticed and define the prognosis factors of a fast evolution.

DETAILED DESCRIPTION:
RATIONAL:

Multiple Myeloma in spite of therapy progresses mainly due to stem cell auto transplant, still remain a deadly disease. About 2000 new cases are diagnosed every year in France. The asymptomatic Stage I MM according to Duries and Salmon's staging are usually only watch over and only treated at progression. Zoledronate is a third generation aminobiphosphonate (BP), probably the most powerful among the available compounds which received market clearance authorisation in MM with bone damage. During MM, bone's hyper resorption is premature. Interactions exist between tumor growth and bone lyses. Zoledronate's got a proper antimyeloma's action (induce plasma cells apoptosis). We propose to test the early use of Zoledronate as soon as stage I MM to delay progression.

STUDY'S OBJECTIVES:

* PRINCIPAL: Assessment of survival without progression stage I MM in two groups: A arm: simple survey and B arm: administration of BP.
* SECONDARY: Describe different progression's type noticed (bone/extra bone) and define the prognosis factor of a fast stage I MM evolution (standard factors, cytogenetic 13 deletion, bone's restructuring strains: crosslaps, bone alkaline phosphatase), list side effects.

STUDY'S KIND:

Multicenter international randomised trial, open labelled, with individual profit.

CONTRIBUTING CENTERS:

Intergroupe Francophone du Myélome's centers.

INCLUSIONS CRITERIA:

Asymptomatic stage I MM without bone's lesion on the standard radiographs.

STUDY'S MONITORING:

After checking inclusion and non inclusion specifications, the patient will be included in the study and randomized (A arm or B arm) before all treatment. The randomisation will be done by center and stratified according to the diagnostic date witch a year or not.

* Arm A: simple survey as standard practice.
* Arm B: a 15 minutes infusion of Zoledronate every month until progression or a maximum of 18 infusions if no progression. The exams are the one usually defined according to good clinical practices guidelines besides cytogenetic, bone's restructuring strain and serum creatin dosage before each infusion in B arm.

STATISTICAL PURPOSES:

The minimum number of patients required showing a median survival time increase without progression of 26 months in the control arm and 38 months in the BP arm is about 175 patients in each arm for a 48 months inclusion's period, and a monitoring of 24 months after the last inclusion (i.e. a study's length of 6 years).

ELIGIBILITY:
Inclusion Criteria:

* stage I multiple myeloma without bones injuries

Exclusion Criteria:

* abnormal kidney function
* VIH infection
* Hepatic incapacity
* pregnancy
* Associate pathology

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 89 (Actual)
Dates: Start 2004-12; Primary Completion 2009-11 (Actual); Study Completion 2012-11 (Actual)

PRIMARY OUTCOMES:
Survival without progress | every month during 6 years

SECONDARY OUTCOMES:
predictive factors of a fast evolution of multiple myeloma | every month during 6 years
Secondary effects of zolédronate | every month during six years

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Gabriel FUZIBET, PU-PH, Principal Investigator — service de médecine interne, CHU de Nice
Locations (1):
- Service de Medecine interne, Hôpital l'ARCHET, CHU de Nice, Nice, France